CLINICAL TRIAL: NCT01598922
Title: Internet Based Cognitive Behavioral Therapy Effects on Depressive Cognitions and Brain Function
Acronym: iCBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Scott Rauch, President and Psychiatrist-in-Chief, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-12-1-0109
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Results first posted 2020-12-07 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Internet Cognitive Behavioral Therapy; fMRI; Neuroimaging
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: For the clinical trial there were only 2 arms: MDD and MAC. There were no Healthy Controls in the CBT vs attention monitoring trial; both groups were depressed.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet Cognitive Behavioral Therapy (Experimental): Participants with major depressive disorder receive an 8-week long internet-based cognitive behavioral therapy program.
  Interventions: Behavioral: Internet Cognitive Behavioral Therapy
- Monitored Attention Control (No Intervention): Participants with major depressive disorder receive no treatment but are monitored closely for 8 weeks. Participants in this arm are offered the treatment at the end of the study.

INTERVENTIONS:
Behavioral: Internet Cognitive Behavioral Therapy — 8 weeks of online treatment program
  Arms: Internet Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to understand the effectiveness of a ten-week internet-based cognitive behavioral therapy (iCBT) treatment on improving depressive symptoms, coping and resilience skills, and cognitive processing.

DETAILED DESCRIPTION:
The need for mental health services is high among military personnel but perceived stigma and other barriers prevent many Soldiers from obtaining the help they need. Alternative mental health treatment approaches that mitigate stigma and increase access and compliance are greatly needed. One promising treatment approach that has shown efficacy in preliminary research and which may address issues related to stigma and barriers to care, is internet-based cognitive behavioral therapy (iCBT). Internet-based treatments offer brief, interactive, and structured treatment approaches that can be completed by individuals relatively anonymously, in the convenience and privacy of their own homes, and according to their own schedules. Such interventions could offer Soldiers an alternative treatment method that minimizes stigma by allowing private and quasi-anonymous access to treatment and which minimizes barriers to care by enhancing access and maximizing schedule flexibility.

Emerging evidence suggests that iCBT is a particularly promising and well-accepted approach for treating large numbers of individuals while minimizing cost and clinicians' time demand. The study of internet-based and other computer-assisted therapies is currently in its infancy and most studies still lack sufficient methodological rigor to firmly establish the efficacy and applicability of these approaches. The proposed project will provide the most comprehensive evaluation of iCBT to date by employing functional neuroimaging techniques, neurocognitive testing of implicit negative biases and responses to negative feedback, and assessment of resilience and coping capacities in addition to standard symptom-based outcome measures.

ELIGIBILITY:
Inclusion criteria:

* Age range between 18 and 45.
* Subjects must be right handed (as measured by Edinburgh Handedness Inventory).
* The primary language of the subjects must be English
* Must have regular access to a computer with internet connection and printer (for potential MDD or MAC participants)
* DSM-IV criteria for current Major Depressive Episode according to SCID (for enrollment into MDD or MAC groups)
* Absence of any psychotropic medications for at least 2 weeks (6 weeks for fluoxetine; 6 months for neuroleptics; 2 weeks for benzodiazepines; 2 weeks for any other antidepressants)
* PHQ-9 score below 5 (for enrollment into HC group)

Exclusion criteria:

* Any history of neurological illness or brain injury
* Current or past DSM-IV Axis I disorder (for enrollment into HC group)
* Complicating medical conditions that may influence the outcome of neuropsychological assessment or functional imaging (e.g., HIV)
* Mixed or left-handedness
* Abnormal visual acuity that is not corrected by contact lenses
* Metal within the body, claustrophobia, or other contraindications for MRI
* Less than 9th grade education
* Past or current alcohol/substance dependence, or current alcohol abuse, or current or past substance abuse (i.e. past alcohol abuse is not exclusionary)
* Use of illicit drugs within the past year
* Use of marijuana within the past month
* Current use of opioid or prescribed stimulant medications
* History of a psychotic mental illness (schizophrenia or bipolar disorder)
* Current severe symptoms of depression (total score > 23 or responding > 1 to Question 9 for suicidal ideation in the Patient Health Questionnaire-9 Item [PHQ-9] (Kroenke et al., 2001))
* A PHQ-9 score below 10 (for potential MDD or MAC participants)
* Currently participating in Cognitive Behavior Therapy
* History of ECT treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Rauch, MD, Principal Investigator — Mclean Hospital
Locations (1):
- Isabelle Rosso, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems, and barriers to care. N Engl J Med. 2004 Jul 1;351(1):13-22. doi: 10.1056/NEJMoa040603. PMID 15229303
- [Background] Titov N, Andrews G, Davies M, McIntyre K, Robinson E, Solley K. Internet treatment for depression: a randomized controlled trial comparing clinician vs. technician assistance. PLoS One. 2010 Jun 8;5(6):e10939. doi: 10.1371/journal.pone.0010939. PMID 20544030
- [Result] Rosso IM, Killgore WD, Olson EA, Webb CA, Fukunaga R, Auerbach RP, Gogel H, Buchholz JL, Rauch SL. Internet-based cognitive behavior therapy for major depressive disorder: A randomized controlled trial. Depress Anxiety. 2017 Mar;34(3):236-245. doi: 10.1002/da.22590. Epub 2016 Dec 23. PMID 28009467
- [Derived] Webb CA, Olson EA, Killgore WDS, Pizzagalli DA, Rauch SL, Rosso IM. Rostral Anterior Cingulate Cortex Morphology Predicts Treatment Response to Internet-Based Cognitive Behavioral Therapy for Depression. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Mar;3(3):255-262. doi: 10.1016/j.bpsc.2017.08.005. Epub 2017 Aug 26. PMID 29486867

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Healthy control subjects were not part of the clinical trial (they were not assigned to treatment).
Groups:
- Internet Cognitive Behavioral Therapy: Participants with major depressive disorder who received a 10-week period of internet-based cognitive behavior therapy (iCBT): 6 online lessons and homework. They also received weekly check-in phone calls, and completed online depression rating scales.
- Monitored Attention Control: Participants with major depressive disorder who received no treatment. These participants logged into the online system the same number of times (6) to complete the same depression self-report scales as participants in the treatment group. They also received the same weekly check-in phone calls as the treatment group during the 10-week period. Participants in this arm were offered the iCBT treatment at the end of the study
Period: Overall Study
Arm/Group | Internet Cognitive Behavioral Therapy | Monitored Attention Control
Started | 37 | 40
Completed | 34 | 30
Not Completed | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Internet Cognitive Behavioral Therapy | Monitored Attention Control | Total
Number analyzed (Participants) | 37 | 40 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (7.7) | 28.8 (6.7) | 29.0 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 53
  Male | 14 | 10 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 23 | 25 | 48
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 6 | 5 | 11
Marital status, married [Count of Participants; unit: Participants] | 5 | 8 | 13
Education [Mean (Standard Deviation); unit: Years] | 15.4 (2.5) | 15.3 (2.0) | 15.4 (2.3)
Employed outside the home [Count of Participants; unit: Participants] | 28 | 24 | 52
Hamilton Rating Scale for Depression, 17 items [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Rating Scale for Depression, 17 item (HRSD-17) was the primary outcome measure of depression severity, administered by doctoral-level raters at pre-treatment/baseline and post-treatment. Each item is rated on a 3- or 5- point scale (0-2 or 0-4), and total HRSD scores can range from 0 to 52. There are 17 items (questions) in this scale, each scored on a 3-point or 5-point scale. Higher scores indicate more severe (worse) symptoms. Total scores vary from 0 to 52. Total scores are represented in this report.
  units on a scale | 15.7 (4.0) | 15.7 (4.3) | 15.7 (4.2)
Patient Health Questionnaire, 9 items [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-9 (PHQ-9) is a well-validated self-report measure of depression severity. The scale presents each of the nine DSM-IV MDD symptoms to be rated on a 4-point frequency scale ranging from "0" (not at all) to "3" (nearly every day). Higher scores indicate more severe (worse) symptoms. Total scores vary from 0 to 27. Total scores are represented in this report.
  units on a scale | 13.9 (3.9) | 15.6 (4.0) | 14.8 (4.0)
Kessler Distress, 10 items [Mean (Standard Deviation); unit: units on a scale] — The Kessler Psychological Distress Scale (K10) is a 10-item self-report measure that yields a score of distress based on questions about anxiety and depressive symptoms that the person has experience in the prior 4 week period. The K10 comprises 10 questions that are answered using a five-point scale (where 5 = all of the time, and 1 = none of the time). The total range of scores is 10 to 50.
  units on a scale | 28.9 (5.4) | 30.8 (4.5) | 29.9 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-treatment to Post-treatment (10 Weeks), Measured by the Hamilton Rating Scale for Depression, 17 Item Version (HRSD-17).
Description: To assess change in severity of depression symptoms. The total score is reported, which is the sum of the ratings of all items and ranges from 0 to 52, with higher scores indicating a worse outcome or greater severity of depression symptoms.
Time Frame: Measured at the baseline visit and 10 weeks after the baseline visit
Population: Note that these are sample sizes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet Cognitive Behavioral Therapy | Monitored Attention Control
Number analyzed (Participants) | 37 | 40
score on a scale
  Pre-treatment HRSD-17 | 15.73 (4.02) | 15.70 (4.26)
  Post-treatment HRSD-17 | 9.17 (6.92) | 14.05 (5.34)
Statistical Analysis 1: Comparison: Internet Cognitive Behavioral Therapy vs Monitored Attention Control; Test type: Other — Intent-to-treat (ITT) analyses following multiple imputation. Generalized Linear Models (GENLIN) predicting post-treatment HRSD scores in the imputed dataset. Covarying for pre-treatment HRSD scores, age and sex; p < 0.0001, GENLIN; Odds Ratio (OR) = 6.11, 95% CI 2-sided [2.814 to 9.403], Standard Error of Mean 1.68

2. Secondary Outcome: Weekly Patient Health Questionnaire (PHQ-9) Score
Description: Participants' scores on the PHQ-9 will be measured at baseline before treatment, each week during the treatment, and again at 10 weeks post-treatment. The range of possible scores on the PHQ-9 is 0 to 27 and higher scores indicate worse outcome or more severe depression
Time Frame: Baseline visit, and 10 weeks after baseline visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Internet Cognitive Behavioral Therapy | Monitored Attention Control
Number analyzed (Participants) | 37 | 40
score on a scale | 9.17 (6.92) | 14.05 (5.34)
Statistical Analysis 1: Comparison: Internet Cognitive Behavioral Therapy vs Monitored Attention Control; Test type: Other; p = .024, hierarchical linear modeling — Hierarchical Linear Modeling (HLM) was applied to PHQ-9 data, adjusting for baseline PHQ-9 score. Group x Time interactions tested for between-group differences in slope of improvement of PHQ-9 scores; Age and sex were covariates. Cohen's d effect sizes are reported; Cohen's d measure of effect size = -0.79, 95% CI 2-sided [-1.25 to -0.32]

3. Secondary Outcome: Weekly Kessler Psychological Distress Scale (K-10) Score
Description: The K-10 is a 10-item self-report measure of psychological distress. Items are scored on a scale from 1" ("none of the time") to "5" ("all of the time"). Total K-10 scores range from 10 to 50, with higher scores reflecting worse outcome or higher distress.
Time Frame: Week 10 score
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet Cognitive Behavioral Therapy | Monitored Attention Control
Number analyzed (Participants) | 37 | 40
units on a scale | 20.14 (7.37) | 26.73 (6.55)
Statistical Analysis 1: Comparison: Internet Cognitive Behavioral Therapy vs Monitored Attention Control; The Kessler Psychological Distress Scale (K-10) is a 10-item scale with total scores that can range from 0 to 50. Higher scores represent worse (more severe) psychological distress; Test type: Other — Hierarchical Linear Modeling (HLM) was applied to K-10 data, adjusting for baseline K-10 score. Group x Time interactions tested for between-group differences in slope of improvement of K-10 scores; p = .003, HLM; Cohen's d measure of effect size = -0.95, 95% CI 2-sided [-1.42 to -0.48]

4. Secondary Outcome: Improvement From Baseline in Brain Functioning on the Emotional Interference Task (EIT) and the Monetary Incentive Delay Task (MID)
Description: At 10 weeks (post-treatment), we will look for improvement from baseline in key brain regions known to be affected by depression. Differences in EIT and MID task-related brain responses will be measured.
Time Frame: baseline, 10 weeks
Population: Analysis still ongoing, anticipated until January 2022
Arm/Group | Internet Cognitive Behavioral Therapy | Monitored Attention Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Positive and Negative Affect Scale (PANAS) Score
Description: Participants' scores on the PANAS will be measured at baseline before treatment, and again at 10 weeks post-treatment. Two scores can be derived. 1) A positive affect score can range from 10 to 50, with higher scores representing better outcome or higher levels of positive affect; 2) Negative Affect score can range from 10 to 50, with higher scores representing better outcome or lower levels of negative affect.
Time Frame: Baseline visit and 10 weeks after baseline visit
Population: Data not analyzed due to funding ending for this study
Arm/Group | Internet Cognitive Behavioral Therapy | Monitored Attention Control
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Connor Davidson Resilience Scale (CD-RISC) Score
Description: Participants' scores on the CD-RISC will be measured at baseline before treatment, and again at 10 weeks post-treatment. Total scores range from 0 to 100, with higher scores indicating a better outcome or higher resilience
Time Frame: Baseline visit, and 10 weeks after baseline visit
Population: Data not analyzed due to funding ending for this study.
Arm/Group | Internet Cognitive Behavioral Therapy | Monitored Attention Control
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Modified Erikson Flanker Test
Description: Participants' scores on the Modified Erikson Flanker Test will be measured at baseline before treatment, and again at 10 weeks post-treatment. Accuracy scores range from 0 to 1 with higher scores reflecting better outcome.
Time Frame: Baseline visit and 10 weeks after baseline visit.
Population: Data still being analyzed and not analysis/paper not anticipated to be completed until January 2022
Arm/Group | Internet Cognitive Behavioral Therapy | Monitored Attention Control
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Implicit Association Test (IAT)
Description: Participants' scores on the IAT will be measured at baseline before treatment, and again at 10 weeks post-treatment. The IAT effect is called the D score with a possible range of -2 to +2, with larger scores reflecting worse outcome and stronger suicidality
Time Frame: Baseline visit, 10 weeks after baseline visit.
Population: Data not analyzed due to funding ending.
Arm/Group | Internet Cognitive Behavioral Therapy | Monitored Attention Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Internet Cognitive Behavioral Therapy | Monitored Attention Control
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/40
Other Adverse Events (participants affected / at risk) | 0/37 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No